CLINICAL TRIAL: NCT04410211
Title: A Comparative Study Between Inhalational Sevoflurane Sedation With Intravenous Midazolam Sedation for Upper Endoscopy Procedure.
Brief Title: Comparison Between Two Types of Sedation for Elective Upper Endoscopy Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Gan Pek Li, Trainee in Anaesthesiology and Critical Care, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2018321-6154
Record Dates: First submitted 2020-05-19; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Gastro Esophageal Reflux; Gastric Ulcer; Sedation Complication
Keywords: Sevoflurane; Midazolam; upper endoscopy; recovery; discharge time
MeSH Terms: conditions — Gastroesophageal Reflux; Stomach Ulcer | interventions — Sevoflurane; Midazolam

STUDY DESIGN:
Intervention Model Description: Patients are randomized to either the Sevoflurane sedation arm or the Midazolam sedation arm based on a randomizer application and the selections are placed in a non-transparent envelope. Once a patient fulfills the eligibility to be recruited in the study, one envelope will be taken to see which arm will the patient be recruited into. Neither the patient nor the investigator will know.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients are randomized to either the Sevoflurane sedation arm or the Midazolam sedation arm based on a randomizer application and the selections are placed in a non-transparent envelope. Once a patient fulfills the eligibility to be recruited in the study, one envelope will be taken to see which arm will the patient be recruited into. Neither the patient nor the investigator will know.
  Two investigators will be selected to participate in this study, whereby one of the investigators who will be providing the care will not be masked. The other investigator who assess the pre and post procedure outcome will be masked from knowing which method is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (inhalational Sevoflurane sedation) (Active Comparator): The inhalational anaesthetic agent and oxygen will be delivered via an anaesthetic circuit with a vaporizer (Sevotec 3, Ohmeda, Streeton UK) with a nasal mask.
  Patients who are allocated for Sevoflurane will be given initial oxygen flow of 8L/min and then Sevoflurane was introduced at a concentration of 0.2% and was increased stepwise by 02% for every 30s up to a maximum of 1.0 minimum alveolar concentration (MAC; 2.05% end tidal). Patient's deepest sedation was recorded and adjusted to achieve optimal Observer's Assessment of Alertness/ Sedation Scale (OAAS) score of 3.
  Inadequate or over sedation was treated by reducing or increasing the Sevoflurane concentration dial by 0.2 - 0.6% until the desired effect is reached.
  Full vital signs monitoring are done for every participant
  Interventions: Drug: Sevoflurane
- Group M (Intravenous Midazolam sedation) (Active Comparator): Patients who are allocated for Midazolam will be given the similar nasal mask delivering 8L/min oxygen. However, Sevoflurane will not be introduced to these patients.
  Midazolam is titrated slowly to achieve OAAS score of 3 but no more than 2.5mg is to be given within 2 minutes period to patients selected to be in Midazolam group.
  Inadequate sedation is treated by giving slow titration of the medication based on the unblinded observer's judgement. Over sedation is treated by withholding the midazolam and continuing oxygen supplementation until the patient returned to the desired sedation level. No other sedative agents are allowed to be given to the patient or else patient will be excluded from this study.
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Sevoflurane — Incidence of side effects such as excitation, headache, apnea, airway obstructions are recorded. Patients who experiences severe excitation disinhibition as defined in the investigator's opinion as agitation. Uncontrollable patient movements that causes unsafe procedural conditions and conversion to general anaesthesia is needed
  Post procedural recovery scoring are taken which includes:
  1. Time taken from the point that the procedure ended to the first OAAS score of 5
  2. Time taken from (a) to meeting discharge eligilibility
  Pre and post procedure pyschometric test (delayed and immediate memory test, posting box test and Stroop test) will be done and compared by the blinded observer/investigator
  Arms: Group S (inhalational Sevoflurane sedation)
Drug: Midazolam injection — Incidence of side effects such as excitation, headache, apnea, airway obstructions are recorded. Patients who experiences severe excitation disinhibition as defined in the investigator's opinion as agitation. Uncontrollable patient movements that causes unsafe procedural conditions and conversion to general anaesthesia is needed
  Post procedural recovery scoring are taken which includes:
  1. Time taken from the point that the procedure ended to the first OAAS score of 5
  2. Time taken from (a) to meeting discharge eligilibility
  Pre and post procedure pyschometric test (delayed and immediate memory test, posting box test and Stroop test) will be done and compared by the blinded observer/investigator.
  Arms: Group M (Intravenous Midazolam sedation)

SUMMARY:
Sedation is defined as the act of administrating a sedative drug to produce a state of calm or sleep. Sedation is commonly given to a patient in hospital settings to provide a tolerable and pleasant experience by relieving anxiety, pain and discomfort, as well as to expedite the duration of the procedure. Moderate sedation (conscious sedation) is the preferred state of sedation, whereby self-maintenance of ventilation and hemodynamic stability is achieved.

The primary objective of this study is to determine if inhalational Sevoflurane is a more superior sedative agent in terms of faster psychomotor recovery and time taken to fulfil discharge criteria when compared with intravenous Midazolam sedation.

Secondary objective is to determine if inhalational Sevoflurane sedation has better patient's and endoscopist's satisfaction when compared with intravenous Midazolam sedation.

DETAILED DESCRIPTION:
A randomized controlled trial study was done on patients undergoing elective upper gastrointestinal endoscopy in a single tertiary Centre in Malaysia. The study was approved by University Malaya Medical Centre medical research ethics committee. All patients gave written and informed consent. Patients were fasted, and three psychometric tests were performed as a baseline before sedation. Patients were randomly allocated to either receive IV Midazolam (Group M) or inhalational Sevoflurane (Group S) via nasal mask. Standard monitoring was applied. Patients in Sevoflurane group received the inhalational agent via a nasal mask with stepwise increment until and Observed Assessment of Alertness/Sedation Scale of 3 or maximum 1.0 minimum alveolar concentration was achieved. Patients in Midazolam group were given a stat dose of IV Midazolam 2.5mg. Both groups received 30mcg of IV Fentanyl and lignocaine 1% gargle prior to the procedure. The unblinded observer monitored the level of sedation and recorded the patient's vital signs. A second blinded observer performed the psychometric tests before and at the end of the procedure. He also recorded the time to fulfil discharge criteria as well as the satisfaction scores from the patient and endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to II
* Patients who are not taking sedative agents prior to procedure.
* Patients who are able to give consent for the procedure.

Exclusion Criteria:

* Patients with ischaemic heart disease, respiratory diseases and cerebrovascular disease.
* Patients who are taking opioid or sedative medications 24 hours before procedure.
* Patients with previous history of adverse effects to Sevoflurane or Midazolam.
* Pregnant patients.
* Patients with airway obstructions.
* Patients with features of difficult airway such as limited neck extension, small mouth opening of less than 3 cm, mallampati score of more than 3.
* Patients who are at risk of aspiration. Impaired gag reflex, presence of neurological disorders and impaired physical mobility.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Psychomotor recovery time | 30 minutes from completion of procedure
  Pre procedure psychomotor tests baseline scores will be obtained and compared with post procedure scores. Time to achieve baseline recovery scores will be taken and used to compare between the two sedative agents.
Time taken to fulfil discharge criteria | One day
  Patient would have to fulfil a set of discharge criteria to ensure that patient is safe for discharge.

SECONDARY OUTCOMES:
Patient and endoscopists satisfaction | Post procedure on the same setting not more than one day duration
  Patient will answer a set of questionnaires to gauge the satisfaction of the sedation agent. Endoscopists will score their satisfaction with a scale of 1 to 10, with 1 - 3 being (dissatisfied), 4-6 (satisfied), and 7 - 10 (very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: PEK LI GAN, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, WP Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after publication

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT04410211/Prot_SAP_ICF_000.pdf